CLINICAL TRIAL: NCT01033279
Title: Evaluation of Self-monitoring of Oral antiCoagulant therApy by the PatiEnts
Brief Title: Quality of Life and Efficacy Evaluation of Patient Self-monitoring Their Oral Anticoagulation Therapy
Acronym: ESCAPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montreal Heart Institute (Other)
Collaborators: Roche Diagnostic Ltd. (Industry)
Responsible Party: Principal Investigator, Lucie Verret, Chief Department of Pharmacy, Montreal Heart Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 09-1158
Record Dates: First submitted 2009-12-15; First posted 2009-12-16 (Estimated); Last update posted 2012-05-30 (Estimated); Status verified 2012-05

CONDITIONS: Anticoagulants; Quality of Life; Drug Monitoring; Pharmacy; Ambulatory Care
Keywords: Coaguchek; Portable coagulometer; Self-monitoring; Coumadin; Warfarin; Quality of life; Pharmacist
MeSH Terms: interventions — Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual care (No Intervention): Patients followed by usual care at the hospital's anticoagulation clinic
- Self-management (Experimental): Self-monitoring and self-adjustment of oral anticoagulation according to predefined algorithms
  Interventions: Other: Self-monitoring and adjustment of oral anticoagulation

INTERVENTIONS:
Other: Self-monitoring and adjustment of oral anticoagulation — Weekly self-monitoring of oral anticoagulation with a portable coagulometer and predefined adjustment algorithms for 4 months following a training program led and designed by hospital pharmacists
  Other Names: warfarin; coumadin; coaguchek XS; coaguchek
  Arms: Self-management

SUMMARY:
The purpose of this study is to determine whether self-management of oral anticoagulation therapy with warfarin has an effect on patient's quality of life following a specific training program led by pharmacists.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years and over followed at the Montreal Heart Institute's Anticoagulation clinic
* Warfarin treatment planned for at least 4 months after inclusion in the study
* Warfarin treatment initiated for at least 6 months
* Last 2 INRs between 1.5 and 4 if target INR is between 2 and 3
* Last 2 INRS between 2 and 4 if target INR is between 2.5 and 3.5
* Provide a signed informed consent

Exclusion Criteria:

* Patient unable to understand (spoken and written) French or English
* Patient refuses or is unable to attend the required training sessions
* Targeted INR other than 2 to 3 or 2.5 to 3.5
* Handicap or physical limitation compromising the patient's ability to initiate self-monitoring in the absence of a proxy helper
* Moderate to severe cognitive impairment or important comprehension problems
* Active neoplasm
* Concurrent chemotherapy
* Hypercoagulable conditions
* Life expectancy of less than 1 year documented in the medical chart
* Inclusion (at time of inclusion or 30 days prior to inclusion) in another research project involving a drug
* Patient anticoagulated with nicoumalone
* Pregnancy or breastfeeding
* Active bleeding (except for menses)
* Recent major bleeding (less than 3 months before inclusion)
* Stroke, acute coronary syndrome, percutaneous coronary intervention, coronary artery bypass graft, cardiac valve replacement, deep veinous thrombosis or pulmonary embolism in the 3 months prior to inclusion
* Any other condition that, in the opinion of the investigators, of the treating physician or of the healthcare professionals working at the anticoagulation clinic could make self-management by the patient impossible

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2009-10; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Anticoagulation-related quality of life | Four months

SECONDARY OUTCOMES:
Time in therapeutic International Normalized Ratio (INR) | Four months
Time in extended therapeutic INR range | Four months
Time in extreme INR ranges (<1.5 and > 5) | Four months
Evolution of anticoagulation-related knowledge post training program | Four months
Time spent by patients managing their oral anticoagulation | Four months
Hemorrhagic events | Four months
Thromboembolic events | Four months

CONTACTS AND LOCATIONS:
Overall Officials: Lucie Verret, B.Pharm, MSc, Principal Investigator — Montreal Heart Institute
Locations (1):
- Montreal Heart Institute, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Verret L, Couturier J, Rozon A, Saudrais-Janecek S, St-Onge A, Nguyen A, Basmadjian A, Tremblay S, Brouillette D, de Denus S. Impact of a pharmacist-led warfarin self-management program on quality of life and anticoagulation control: a randomized trial. Pharmacotherapy. 2012 Oct;32(10):871-9. doi: 10.1002/j.1875-9114.2012.01116. PMID 23033226